CLINICAL TRIAL: NCT02222701
Title: Composite Resins Reconditioned, Behavior and Survival: Clinical Follow-up 10 Years
Acronym: reacondcomp
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Eduardo Fernandez Godoy, University of Chile
Other Study IDs: FOUCH2012/10-4
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Unsatisfactory Restoration of Tooth
Keywords: composite; dental; longevity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Replacement: Composite resins with Alpha values for the marginal adaptation criteria were used as the positive control and were made with resin composite (Filtek Supreme, 3M ESPE), eith rubber dam isolation and the adhesive system L-Pop Prompt (3M-ESPE)
- No treatment: Composite resin restorations (Z100, 3M ESPE) in general clinically acceptable, did not receive treatment.
- Refurbishing: For this group, The dentists finished the occlusal, lingual or facial surfaces of defective RBC restorations with the medium series of aluminum oxide disks (Sof-Lex,3M ESPE) or carbide burs (12 and 30 blades,Brasseler USA, Dental Instrumentation,Savannah, Ga.) and then polished them with afine series of aluminum oxide disks (Sof-Lex, 3M ESPE) and diamond-impregnated composite polisher (ComposiPro Diacomp, Brasseler). For restorations in which proximal surface areas were affected, the clinicians smoothed them with interproximal aluminum oxide finishing strips (Sof-Lex Finishing Strips, 3M ESPE).

SUMMARY:
The purpose of this study is to evaluate the clinical performance of resin composite restorations refurbished and compare with 2 groups of resins, 1 without treatment and another replaced resins acted as controls. The null hypothesis of this study is that the group of refurbished resins have a similar behavior to the control groups.

DETAILED DESCRIPTION:
A cohort of 26 patients aged 18-80 years old (mean: 28.35 years; 42% men, 58% women) with 78 composite restorations (Class I: 39; Class II: 39) were recruited at the Operative Dentistry Clinic at the Dental School of the University of Chile. All participants in the refurbishing groups showed clinical features for the anantomy, roughness and/or luster that deviated from the ideal and were rated Bravo according to the modified United States Public Health Service (USPHS) criteria. New Composites with Alpha values (Replacement group) and acceptable composites (No treatment group) were used as controls. The protocol was approved by the Institutional Research Ethics Committee of the Dental School at the University of Chile (Project PRI-ODO-0207). All patients signed informed-consent forms and completed registration forms

General Inclusion Criteria:

* Patients with more than 20 teeth.
* Restorations in functional occlusion, with an opposing natural tooth.
* Asymptomatic restored tooth.
* At least one proximal contact area with a neighboring tooth.
* Patients older than 18 years.
* Patients who agreed and signed a consent form for participating in the study.
* Area outside of the restoration failure is in good condition.

General Exclusion Criteria:

* Patients with contra-indications for regular dental treatment based on their medical history.
* Patients with xerostomia or individuals taking medication that significantly decreased salivary flow.
* Patients with a high risk of caries.
* Patients with psychiatric or physical diseases, which interfered with oral hygiene.

Treatment Group Criteria Two hundred four patients were initially evaluated and assigned in accordance with the modified USPHS criteria,26 patients were selected based on the inclusion criteria with at least 1 Composite restoration with anatomy, roughness and/or luster (Bravo) suitable for reburbishing, with another composite restorations that had excellent values (Alpha) and was made at this time (Replacement group).And finally another composite pre-existing with acceptable condition (Alpha or Bravo values) acted as control. The patient was considered the statistical unit in this study (n=20).

Restoration Assessment The quality of the restorations was scored in accordance with the modified USPHS criteria. The Cohen Kappa inter-examiner coefficient was 0.74 in the first year and 0.87 after 10 years for two examiners (JM and EF) who underwent calibration training exercises each year. In the first, second, third, fourth, fifth, and tenth years, the examiners independently assessed the restorations for anatomic form, roughness, color, marginal staining,luster, secondary caries, marginal and marginal adaptation, both directly via tactile and visual examinations with mouth mirror number five and explorer number 23 (Hu Friedy Mfg. Co. Inc.) and indirectly by radiographic examination (bite wing). A third clinician (GM), who also underwent the calibration training exercises, made the final decision if a difference was recorded between the two examiners and they could not reach an agreement.

Treatment Groups Refurbishing For this group, The dentists finished the occlusal, lingual or facial surfaces of defective RBC restorations with the medium series of aluminum oxide disks (Sof-Lex,3M ESPE) or carbide burs (12 and 30 blades,Brasseler USA, Dental Instrumentation,Savannah, Ga.) and then polished them with afine series of aluminum oxide disks (Sof-Lex, 3M ESPE) and diamond-impregnated composite polisher (ComposiPro Diacomp, Brasseler). For restorations in which proximal surface areas were affected, the clinicians smoothed them with interproximal aluminum oxide finishing strips (Sof-Lex Finishing Strips, 3M ESPE).

Replacement group Composite resins with Alpha values for the marginal adaptation criteria were used as the positive control and were made with resin composite (Filtek Supreme, 3M ESPE), eith rubber dam isolation and the adhesive system L-Pop Prompt (3M-ESPE) No treatment Composite resin restorations (Z100, 3M ESPE) in general clinically acceptable, did not receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 20 teeth.
* Restorations in functional occlusion, with an opposing natural tooth.
* Asymptomatic restored tooth.
* At least one proximal contact area with a neighboring tooth.
* Patients older than 18 years.
* Patients who agreed and signed a consent form for participating in the study.
* Area outside of the restoration failure is in good condition.

Exclusion Criteria:

* Patients with contra-indications for regular dental treatment based on their medical history.
* Patients with xerostomia or individuals taking medication that significantly decreased salivary flow.
* Patients with a high risk of caries.
* Patients with psychiatric or physical diseases, which interfered with oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any person with composite restorations
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2003-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in quality of restorations | 1 year
  The quality of the restorations was scored according to the modified USPHS criteria. Two examiners underwent calibration exercises each year (JM and EF). Immediately after the treatment (baseline) and 10 years later, the examiners assessed the restorations independently by direct visual and tactile examination with mouth mirror number 5 and explorer number 23 (Hu Friedy Mfg. Co. Inc., Chicago, IL, USA) and indirectly by radiographic examination (bite wing). The four parameters examined were anatomic form, secondary caries, marginal staining and marginal adaptation. If the difference was recorded between the two examiners, and if they could not reach an agreement, a third clinician, who also underwent the calibration exercises (GM), made the final decision.

CONTACTS AND LOCATIONS:
Overall Officials: eduardo fernandez, Principal Investigator — University of Chile
Locations (1):
- Eduardo Fernandez Godoy, Santiago, Chile

REFERENCES:
- [Result] Moncada G, Vildosola P, Fernandez E, Estay J, de Oliveira Junior OB, de Andrade MF, Martin J, Mjor IA, Gordan VV. Longitudinal results of a 10-year clinical trial of repair of amalgam restorations. Oper Dent. 2015 Jan-Feb;40(1):34-43. doi: 10.2341/14-045-C. Epub 2014 Aug 6. PMID 25100406
- [Result] Fernandez E, Martin J, Vildosola P, Oliveira Junior OB, Gordan V, Mjor I, Bersezio C, Estay J, de Andrade MF, Moncada G. Can repair increase the longevity of composite resins? Results of a 10-year clinical trial. J Dent. 2015 Feb;43(2):279-86. doi: 10.1016/j.jdent.2014.05.015. Epub 2014 Jun 4. PMID 24907560